CLINICAL TRIAL: NCT03076788
Title: Intracardiac Flow Remodeling in Athletes
Acronym: INFINITE
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Amir HODZIC, Medical Doctor, University Hospital, Caen
Other Study IDs: 16-022.
Record Dates: First submitted 2017-02-16; First posted 2017-03-10 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Remodeling, Ventricular
Keywords: echocardiography; intraventricular pressure gradients; cardiac remodeling; athletes
MeSH Terms: conditions — Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Athletes: Professional and amateur athletes examined during the medical follow-up at the medical sport centre of Caen University Hospital.
  The medical examination consists in a clinical exam, an electrocardiogram and an echocardiography.
  Interventions: Other: electrocardiogram and echocardiography
- Sedentary controls: Sedentary patients assessed in the cardiology unit with a normal heart function.
  The medical examination consists in a clinical exam, an electrocardiogram and an echocardiography.
  Interventions: Other: electrocardiogram and echocardiography

INTERVENTIONS:
Other: electrocardiogram and echocardiography — We retrieved all electrocardiograms and echocardiography made during the clinical examination of each athlete and each sedentary control.
  * Standard 12 lead ECG
  * Trans-thoracic echocardiography examination of cardiac function, morphology and intracardiac flow.

SUMMARY:
The uncertainty concerning the onset and the extent of cardiac remodeling in response to intensive training hinders medical evaluation by physician. A better knowledge of the physiology of cardiac adaptation to training will enable physicians to correctly determine whether observed patterns of cardiac remodeling are physiological or pathological. This prospective study proposes to assess in a trained-athlete population the cardiac remodeling in response to intensive exercise training. This study is observational, we do not interfere with athlete's training.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18yrs old
* Ability to give written consent for participating in the study

Exclusion Criteria:

* Age < 18yrs old
* Cardiac diseases, arterial hypertension, cardiac devices, diabetes, renal, liver or pulmonary failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Athletes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of ventricular response to exercise training by echocardiography. | Day 1
  1. 2D- morphological and functional parameters of both left and right ventricles:
     * end-diastolic and end-systolic dimensions (cm)
     * left ventricular mass (g)
     * ventricular end-diastolic and end-systolic areas (cm²)
     * ventricular ejection fraction (%)
     * atrial volumes (ml)
     * diastolic indices by pulsed wave Doppler and tissue Doppler (cm/s)
     * myocardial deformation by speckle tracking (%)
  2. 3D- morphological and functional parameters of both left and right ventricles:
     * ventricular full volumes (ml)
     * ejection fraction (%)
  3. Intracardiac flow measurements by color Doppler M-mode:
  estimation of intra ventricular pressure gradients between the base and the apex (mmHg).

SECONDARY OUTCOMES:
Evaluation of ventricular response to exercise training by electrocardiogram | Day 1
  * heart rate (bpm),
  * ventricular hypertrophy (mV)
  * atrial remodeling (mV)
Sport and medical history questionnaire | Day 1
  exercise training program, medical past history, cardiovascular risk factors, treatments, doping.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de CAEN, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No